CLINICAL TRIAL: NCT00432887
Title: Caffeine and Glucose Regulation
Brief Title: Experimental Studies of the Effects of Caffeine on Glucose Regulation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DK67486 (completed)
Record Dates: First submitted 2007-02-05; First posted 2007-02-08 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: caffeine; coffee; glucose; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

INTERVENTIONS:
Drug: caffeine administration

SUMMARY:
This project contains experimental studies of the effects of the drug caffeine on glucose regulation in adults who have Type 2 diabetes. In our experiments, we are testing the hypothesis that moderate amounts of caffeine exaggerate the abnormal increases in glucose and insulin observed after meals in patients with type 2 diabetes. On separate study days subjects receive standard meals after taking capsules containing either caffeine or an inactive placebo. We measure levels of glucose, insulin, and other chemicals in blood samples drawn over the next 3 hours. In a separate study, we use continuous glucose monitoring to measure glucose levels during everyday activities on days when subjects receive caffeine or placebo.

These studies do not involve clinical treatment or disease management. However, we hope to learn whether a very popular drug impairs the clinical management of a common disease.

DETAILED DESCRIPTION:
Pilot results suggest that caffeine, the most commonly used drug in the world, may interfere with postprandial glucose metabolism by increasing insulin resistance and/or by stimulating hepatic glucose production. This effect could have serious clinical implications for coffee drinkers who have type 2 diabetes. Early results suggest caffeine exaggerates the postprandial hyperglycemia and hyperinsulinemia present in these patients.

The experimental (non-treatment) studies in this project include double-blind placebo-controlled cross-over laboratory tests of glucose tolerance in groups of type 2 diabetic patients and prediabetic volunteers who are coffee drinkers.

The lab studies test the hypothesis that caffeine (vs. placebo) increases postprandial insulin responses and results in a potentiation of glucose responses in the type 2 group.

An ambulatory study examines the effects of caffeine administration on glucose levels during everyday activities in the natural environment. This study uses a double-blind placebo-controlled cross-over design. Ambulatory glucose data are collected with a MiniMed CGMS sensor and recorder worn for 72 hours. Caffeine and placebo are administered on separate days. Average glucose levels and glucose responses to meals are compared across treatment days within subjects.

ELIGIBILITY:
Inclusion criteria:

* 6 months or longer history of type 2 diabetes
* treatment by diet, exercise, or oral medication
* current daily consumption of 2 or more cups of coffee
* BMI >21kg/M2 and < 45kg/M2

Exclusion criteria:

* Required use of insulin
* Current cigarette smoking
* Current use of medications that impact glucose metabolism
* Pregnancy
* Other major medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-07; Study Completion 2007-02

PRIMARY OUTCOMES:
postprandial glucose and insulin
fasting glucose and insulin
insulin resistance
glucose tolerance

SECONDARY OUTCOMES:
epinephrine
norepinephrine
cortisol
blood pressure
plasma caffeine concentration

CONTACTS AND LOCATIONS:
Overall Officials: James D. Lane, Ph.D., Principal Investigator — Duke University